CLINICAL TRIAL: NCT05355948
Title: A Prospective, Multi-Center, Randomized Clinical Trial to Evaluate the Detection of Atrial Fibrillation for an One Day Versus More Than or Equal to Eight Days Using MEMO Patch PLUS in Individuals Aged ≥ 75 Years, or Those at High Risk of Stroke: MEMO-DAF8
Brief Title: A Clinical Trial to Evaluate the Detection of Atrial Fibrillation for an One Day Versus More Than or Equal to Eight Days Using MEMO Patch PLUS in Individuals Aged ≥ 75 Years, or Those at High Risk of Stroke
Acronym: MEMO-DAF8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-2022-0008
Record Dates: First submitted 2022-04-21; First posted 2022-05-02 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation/Flutter in Patients With High Risk of Stroke
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEMO Patch PLUS ECG monitoring for One-day (Experimental)
  Interventions: Device: MEMO Patch PLUS for 1 day
- MEMO Patch PLUS ECG monitoring for More than 8-days (Experimental)
  Interventions: Device: MEMO Patch PLUS for More than 8-days

INTERVENTIONS:
Device: MEMO Patch PLUS for 1 day — Individuals randomized to one-day monitoring will wear MEMO Patch PLUS for 1 day. After that, confirm the monitoring result and carry out a fixed schedule.
  Arms: MEMO Patch PLUS ECG monitoring for One-day
Device: MEMO Patch PLUS for More than 8-days — Individuals randomized to More than 8-days monitoring will wear MEMO Patch PLUS for 8 days ~ 14 days at their voluntarily. After that, confirm the monitoring result and carry out a fixed schedule.
  Arms: MEMO Patch PLUS ECG monitoring for More than 8-days

SUMMARY:
The purpose of this study is to evaluate the benefits in the atrial fibrillation detection rate of the continuous ECG monitoring group for more than 8 days by contrasting with one-day ECG monitoring using MEMO Patch PLUS in 1000 patients with atrial fibrillation-related symptoms in the high risk group of stroke. The participant is allocated randomly to One-day ECG monitoring group or the continuous ECG monitoring group for more than 8 days in ratio of 1:1, only if the participant provides informed consent and eligible for all the inclusion/exclusion criteria. The investigator confirms the results of MEMO Patch PLUS monitoring at 1 month from the date of MEMO Patch PLUS attachment. The participation of the subject is terminated on the 1 year from the date of MEMO Patch PLUS attachment. On that day, investigator evaluates incidence of the event associated with atrial fibrillation, the event is included ischemic stroke/transient ischemic accident, hemorrhagic stroke, systemic embolism, etc.

ELIGIBILITY:
[Inclusion criteria]

A participant will be eligible for inclusion in the study if the participant:

1. Has provided documented informed consent for the study.
2. Is adult at least 19 years of age on the day of providing documented informed consent
3. Is the high risk group for stroke, i.e. adult at least 75 years of age or CHA2DS2-VASc score more than 2
4. Is life expectancy more than 6 months
5. Has no Atrial fibrillation or Atrial flutter as a result of 12-lead ECG
6. Has symptoms associated with Atrial fibrillation *symptoms associated with Atrial fibrillation: palpitation, dizziness, dyspnea, syncope, stroke/transient ischemic accident, systemic embolism etc.

[Exclusion criteria]

The participant must be excluded from the study if the participant:

1. Has had prior history of Atrial fibrillation or Atrial flutter
2. Has received prior or ongoing anticoagulant or antiplatelet therapy
3. Has inserted Pacemaker or Defibrillator that can diagnose Atrial fibrillation or Atrial flutter
4. Has plan of Carotid endarterectomy or inserting Stent* within 90 days on the day of providing document informed consent *Stent insertion: means when stent-related interventions have been performed on the carotid arteyr or coronary arteries.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of newly diagnosed AF | 1 month(+1month)
  Incidence of newly diagnosed AF refers to a case that lasts longer than 30 seconds, which is an indication for anticoagulation or antiplatelet therapy in standard therapy.
Incidence of newly diagnosed AF | 2 month(±Month 2)
  Incidence of newly diagnosed AF refers to a case that lasts longer than 30 seconds, which is an indication for anticoagulation or antiplatelet therapy in standard therapy.

SECONDARY OUTCOMES:
Time to the first occurrence of atrial fibrillation/flutter lasting more than 30 seconds after MEMO Patch PLUS is attached. | 1month(+1month), 12 month(±Month 2)
Adaptation rate of anticoagulant or antiplatelet therapy when atrial fibrillation/flutter is diagnosed. | 1month(+1month), 12 month(±Month 2)
Time required to use or switch to anticoagulant or antiplatelet therapy after atrial fibrillation/flutter diagnosis. | 1month(+1month), 12 month(±Month 2)
Burden of total atrial fibrillation/flutter occurrence time | 1month(+1month), 12 month(±Month 2)
Incidence of significant medical events or death due to ischemic stroke/transient ischemic attack, systemic embolism, hemorrhagic stroke, atrial fibrillation/flutter. | 1month(+1month), 12 month(±Month 2)
Percentage of arrhythmias including atrial fibrillation/flutter were detected and surgery/procedure was performed for therapeutic or diagnostic purposes. | 1month(+1month), 12 month(±Month 2)
Distribution rate of wearing period of ECG monitoring group for more than 8 days. | 1month(+1month), 12 month(±Month 2)
Detection rate of other arrhythmias* except atrial fibrillation/flutter. | 1month(+1month), 12 month(±Month 2)

CONTACTS AND LOCATIONS:
Overall Officials: Boyoung Joung, Principal Investigator — Severance Cardiovascular Hospital Yonsei University
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park SH, Jin JH, Kim J, Lee D, Kim D, Jang J, Yu HT, You SC, Joung B. Wearable device derived electrocardiographic age and its association with atrial fibrillation. NPJ Digit Med. 2026 Jan 17. doi: 10.1038/s41746-026-02344-8. Online ahead of print. PMID 41548032